CLINICAL TRIAL: NCT06461260
Title: Safety, Efficacy and Neuroimaging Mechanisms of Amygdala Temporal Interference Stimulation Therapy for Depression
Brief Title: Amygdala MRI-TIS for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pudong New Area Mental Health Center, School of Medicine, Tongji University (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jingjing Huang, MD, Chief Physician, Shanghai Pudong New Area Mental Health Center, School of Medicine, Tongji University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDJW-2024-001CSA
Record Dates: First submitted 2024-05-31; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Deep Brain Stimulation; TI stimulation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amygdala TI (Experimental): Right amygdala Temporal Interference (TI) stimulation with 100 frequency difference, 20 minutes per day for 5 days.
  Interventions: Device: Nervio-X

INTERVENTIONS:
Device: Nervio-X — An 8-channel TIS device developed by NEURODOME Corporation.

SUMMARY:
The study utilizes a non-invasive deep brain stimulation (temporal interference, TI) technique primarily targeting the amygdala to preliminarily explore the clinical efficacy and potential mechanisms of MRI-compatible TI technology in regulating the amygdala in depressive disorders, providing a more comprehensive basis for the application of TI technology.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged between 18 and 65, with no gender restrictions;
* A diagnosis of depression made by the study physician based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
* HAMD-17 score of 17 or higher;
* Participants must not have changed their antidepressant medication regimen from 30 days prior to signing the informed consent form through the duration of the experiment;
* Eligible individuals or their authorized representatives must demonstrate, as assessed by the study physician, a comprehensive understanding of the study's objectives and procedures, be capable of adhering to the requirements set forth in the study protocol, and provide their signature on the informed consent form.

Exclusion Criteria:

* Eligible participants must not have a history of psychiatric or neurological disorders, as judged by the investigator, which may impact the evaluation of the study's efficacy;
* Participants must not have a history of seizures or prior episodes of epilepsy;
* The presence of metallic foreign objects within the cranial structure or metallic cardiac implants;
* Participants must not have a diagnosis of organic brain disease, nor a history of significant cranial trauma or neurosurgical intervention;
* Participants received electroconvulsive therapy or other physical therapies (such as transcranial magnetic stimulation therapy);
* The researcher evaluated the individual's mental state and determined it to present a significant risk of suicidal ideation or behavior;
* Pregnant or breastfeeding;
* Participants who are concurrently engaged in other clinical interventional trials;
* Participants presenting with other circumstances that the investigator deems unsuitable for the intervention being studied

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
HAMD-17 | Baseline, treatment completion day, 1 week, 4 weeks and 8 weeks

SECONDARY OUTCOMES:
HAMA | Baseline, treatment completion day, 1 week, 4 weeks and 8 weeks
  HAMA is a questionnaire that designed to evaluate the presence and intensity of anxiety symptoms in both clinical and research settings.
SHAPS | Baseline, 4 weeks and 8 weeks
  The SHAPS is a questionnaire that used to measure the severity of anhedonia, a common symptom in various mental health conditions.
SF-36 | Baseline and 8 weeks
WHOQOL-BREF | Baseline and 8 weeks
PSQI | Baseline, 4 weeks and 8 weeks
THINC-it® | Baseline, treatment completion day and 8 weeks
  THINC-it® is a screening tool for assessment of cognitive functioning in patients with a major depressive episode/disorder
Blood sample | Baseline, 4 weeks
  Peripheral blood will be collected at baseline and one 4 weeks after treatment for transcriptomic and proteomic studies to explore the molecular mechanisms of temporal interference (TI) in the treatment of depressive disorders and to identify molecular markers for predicting therapeutic efficacy
GAD-7 | Baseline, treatment completion day, 1 week, 4 weeks and 8 weeks
QIDS-SR | Baseline, treatment completion day, 1 week, 4 weeks and 8 weeks
MADRS | Baseline, treatment completion day, 1 week, 4 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pudong New Area Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No